CLINICAL TRIAL: NCT03139422
Title: Tranexamic Acid Versus Calcium Dobesilate for the Treatment of Copper Intra Uterine Contraceptive Device Associated Heavy Menstrual Blood Loss : A Randomized , Open-labelled , Clinical Trial.
Brief Title: Treatment of Copper Intra Uterine Device Associated Heavy Menstrual Blood Loss
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TA
Record Dates: First submitted 2017-04-30; First posted 2017-05-04 (Actual); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Menorrhagia
MeSH Terms: conditions — Menorrhagia | interventions — Tranexamic Acid; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tranexamic Acid (Active Comparator): Tranexamic Acid oral tablets 500 mg every six hour with the onset of the first day of menstrual cycle till the end of bleeding for 3 cycles
  Interventions: Drug: Tranexamic Acid 500 MG
- Calcium Dobesilate (Experimental): Calcium Dobesilate oral tablets 500 mg (three times daily) with the onset of the first day of menstrual cycle till the end of bleeding.
  Interventions: Drug: Calcium Dobesilate

INTERVENTIONS:
Drug: Tranexamic Acid 500 MG — oral tablets
  Arms: Tranexamic Acid
Drug: Calcium Dobesilate — oral tablets
  Arms: Calcium Dobesilate

SUMMARY:
Intrauterine contraceptive device is the most commonly reversible method used among women of reproductive age worldwide. Almost one in five married contraceptive users is currently using Intrauterine contraceptive device. The Egyptian demographic and health survey results indicate that 30% of currently married women interviewed in the Egyptian demographic and health survey were using Intrauterine contraceptive device. Main reasons for discontinuation of Intrauterine contraceptive device as cited by women were excessive bleeding per vagina 39.68%, abdominal pain 38.62%, low backache35.97%.

ELIGIBILITY:
Inclusion Criteria:

1. Women usingsopperT380A and reporting heavy menstrual blood loss during use.
2. Menorrhagia , will be defined as a Pictorial blood loss assessment chart-Score greater than 100.
3. No contraindication to drugs used in treatment.
4. No other cause for heavy menstrual blood loss

Exclusion Criteria:

1. Refusing to participate.
2. Irregular menstrual cycle.
3. Misplaced Intrauterine device.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-10 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Percent of women requesting treatment for heavy menstrual blood loss. | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut Faculty of Medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No